CLINICAL TRIAL: NCT06678113
Title: A Phase 1b, Single Arm, Multi-center, Open-label, Dose-escalation Study to Assess the Safety and Efficacy of Intravenous BSG005 in Patients With Invasive Fungal Infection
Brief Title: Study to Assess the Safety and Efficacy of Intravenous BSG005 in Patients With Invasive Fungal Infection
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Biosergen AS (Industry)
Collaborators: Alkem Laboratories Ltd (Industry); JSS Medical Research Asia pacific Private Limited (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BSG-1.02
Record Dates: First submitted 2024-08-29; First posted 2024-11-07 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2024-08

CONDITIONS: Invasive Fungal Infection
Keywords: Invasive fungal infection; BSG005; Polyene macrolide; Rescue therapy
MeSH Terms: conditions — Invasive Fungal Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Active treatment (Experimental): The patient will receive active treatment in a dose escalation manner increasing the dose every 3 days dependent on safety and efficacy
  Interventions: Drug: BSG005

INTERVENTIONS:
Drug: BSG005 — Single arm dose escalation in patients with invasive fungal infection
  Other Names: Polyene Macrolide

SUMMARY:
This study is an open-label, Phase 1b, dose-escalation/finding study to assess the safety and efficacy of intravenous BSG005 in patients with uncomplicated invasive fungal infections (IFI).

Approximately 15 patients are planned to be enrolled in 3 cohorts. The study will be conducted in 3 cohorts consisting of 3 periods, namely: Screening, Treatment, and Follow-up periods. In each cohort, 5 patients are planned to be enrolled.

This study is a single-arm study. The treatment (BSG005) in each dose level will be administered once daily for 3 days via IV infusion. If the safety and tolerability profiles are acceptable at each dose level, the patients will be treated for a maximum of 28 days. Each patient will be in the study for up to 50 days, which consists of a 7-day Screening period, 1 day for baseline assessments, up to 28 days (maximum) of treatment with BSG005, and 14 days of follow-up.

DETAILED DESCRIPTION:
This study is an open-label, Phase 1b, dose-escalation/finding study to assess safety and efficacy of intravenous BSG005 in patients with uncomplicated invasive fungal infections (IFI).

The study will be conducted in 3 cohorts consisting of 3 periods, namely: Screening, Treatment, and Follow-up periods. In each cohort, 5 patients are planned to be enrolled. Following 7 days of Screening period, patients will be enrolled in the study. In Cohort 1, patients will be administered with a dose of 0.1 mg/kg, which was tested in the single ascending dose (SAD) group of the Phase 1 healthy subject study and will follow an intra-patient dose-escalation step. Based on the overall health status of the patient (safety and efficacy of study intervention), the dose can be adjusted at any point of time according to the Investigator´s judgment, which would be based on clinical or mycological or radiological assessments dependent on the information available. This can be dose escalation or dose de-escalation as appropriate. During the Treatment period, there may be a pause of one day or more if deemed necessary by the Investigator. Each patient will be evaluated individually for efficacy and safety to decide if escalation is possible. The dose will be escalated by 0.1 mg/kg every 3 days or 1 day earlier (ie, 2 days) at the Investigator's discretion.

The starting dose in Cohort 1 will be 0.1 mg/kg for the first 3 days of treatment; if no safety concerns are experienced, the patients will be escalated up to 0.2 mg/kg. This process will be followed up to a maximum of 1.0 mg/kg or till a maximum of 28 days of treatment duration in Cohort 1, with the possibility to stop anytime after 14 days depending on the status of the patient. The starting dose of Cohort 2 will be decided by the Data Safety Review Committee (DSRC) after review of all available relevant data up to Day 14 of treatment for all patients in Cohort 1. Subsequently, a similar dose-escalation will be followed for Cohort 2 as defined above for Cohort 1. The dose can be escalated up to a maximum of 2.0 kg/mg. A similar process will be followed for the first dose in Cohort 3 and the dose can be escalated up to a maximum of 3.0 mg/kg. BSG005 will be administered daily via IV infusion for 120 minutes (may be prolonged for up to 240 minutes). As BSG005 has a propensity for phlebitis, central catheters or long peripheral catheters are preferred for infusion.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years.
2. Able to provide written informed consent or have a legally authorized representative that can provide informed consent in case of incapacitation.
3. Diagnosed by Investigator to have an IFI.

   - Proven IFIs as defined in the 2020 consensus definitions by the European Organization for Research and Treatment of Cancer/ Mycoses Study Group Education and Research Consortium (EORTC/MSGERC). Probable or possible IFIs can be included using the EORTC/MSGERC criteria or other established criteria. The inclusion of patients with IFI caused by, eg, Aspergillus spp and Candida spp, is preferred as these species are generally known to be responsive to a lower dose than other species, eg, Mucor mycosis
4. IFI patients with mild to moderate renal impairment or IFI patients requiring an alternative treatment as current treatment cannot be continued due to any of the following

   1. Failure with one first-line agent, defined as either: Radiologic progression, Increase in serologic markers such as galactomannan antigen or beta-D-glucan, Failure of clearance of cultures , Progression or lack of improvement in a clinically appropriate timeframe of clinical symptoms attributed to IFI;
   2. Inability to tolerate AmB, as defined by at least one of the following: Nephrotoxicity with either: 1.5 mg/dL increase in creatinine from baseline, 50% increase in creatinine from baseline ii. Contraindication to use AmB with either:- Persistent hypokalemia or hypomagnesemia while on AmB despite appropriate electrolyte replacement
   3. Documented in vitro resistance to first-line antifungal therapy (ie fluconazole resistance in Candida auris)
   4. Treatment-limiting drug-drug interactions prohibiting the use of antifungals (azoles and echinocandins) such as concurrent rifampcin, rifabutin, phenytoin, carbamazepine, bedaqualine

Exclusion Criteria:

1. Patient has a known hypersensitivity or severe infusion-related reaction to any polyene drug.
2. Infection caused by a known or suspected organism with intrinsic resistance to AmB.
3. Concurrent use of another investigational agent within 30 days of enrollment.
4. Chronic kidney disease with estimated glomerular filtration rate (eGFR) less than 30 mL/min or dialysis. Patients with acute kidney injury with eGFR less than 30 mL/min and improving creatinine level can be included as judged by the Investigator.

   Note: Patients may be rescreened within 48 hours if laboratory values are found to be abnormal.
5. Has liver enzyme results (aspartate aminotransferase [AST]/alanine aminotransferase [ALT]) greater than 5 times the upper limit of normal.

   Note: Patients may be rescreened within 48 hours if laboratory values are found to be abnormal.
6. Has a bilirubin level greater than 5 times the upper limit of normal. Note: Patients may be rescreened within 48 hours if laboratory values are found to be abnormal.
7. Patients who have an ejection fraction less than 25% of predicted.
8. Currently pregnant or planning on getting pregnant while on study (details of contraception guidance are provided in Section 13).
9. Breastfeeding.
10. Patients not likely to survive a minimum of 28 days from start of screening.
11. Patient receiving prohibited medications.
12. Patient is an abuser of alcohol or medication.

    -

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
To establish the safety and tolerability of BSG005 in patients with severe invasive fungal infection | From enrollment to end of treamtent including 14 days follow up
  Treatment Emergent Adverse Event (CTC grading of severity)
To establish the safety and tolerability of BSG005 in patients with severe invasive fungal infection | From enrollment to end of treamtent including 14 days follow up
  Renal function (eGFR)

SECONDARY OUTCOMES:
To assess the overall response to BSG005 treatment in patients with invasive fungal infection | From treatment start to end of treatment plus 14 days follow up
  Overall response as per guidelines (composite of clinical, radiology, microbiology) Treatment success - complete & partial response, & stabile disease Treatment failure - progression Dose estimation for treatment success based on fungal infection strain Mortality during the course of the study (crude & associated)
To assess the overall response to BSG005 treatment in patients with invasive fungal | From treatment start to end of treatment plus 14 days follow up
  To guide dose selection for future testing

CONTACTS AND LOCATIONS:
Overall Officials: Tine Olesen, PhD, Study Chair — BIOSERGEN AB
Locations (1):
- JSS Medical Research Asia Pacific Private Limited, Dehli, Haryana, India

IPD SHARING:
Plan to Share IPD: Yes
Safety and efficacy data will be shared
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The information will be available after end of study when the clinical trial report is written
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information or to submit a request, please contact tine.olesen@biosergen.net
URL: https://www.biosergen.net/